CLINICAL TRIAL: NCT01479777
Title: FES Driven Stepping in Individuals With Spinal Cord Injury
Brief Title: Functional Electrical Stimulation (FES) Driven Stepping in Individuals With Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Cristina Sadowsky, M.D., Assistant Professor Physical Medicine and Rehabilitation, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00016421
Record Dates: First submitted 2011-11-15; First posted 2011-11-24 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2014-09-15 (Estimated); Status verified 2014-09

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury; Functional electrical stimulation; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FES Stepping (Experimental): For the next 8 weeks, we will ask you to come to the ICSCI twice (2) time per week during which you will perform FES Stepping.
  Interventions: Device: FES Stepping (RT600 from Restorative Therapies, INC.)

INTERVENTIONS:
Device: FES Stepping (RT600 from Restorative Therapies, INC.) — You will be transferred to the RT600 device and secured in a support harness. We will place your legs onto the RT600 device and secure them with straps. Electrodes (pads that stick to the skin) will be placed on your skin on your legs, buttock, stomach, and back. The pads will be connected to a stimulator box through a wire. We will then start the stepping motor and stimulate your muscles with electric current. This will cause your legs to step. You will do this for 1 hour.
  Other Names: RT600 from Restorative Therapies, INC.

SUMMARY:
The research is being done to find out if Functional Electrical Stimulation (FES) stepping can improve the function of people with spinal cord injury that paralyzes.

DETAILED DESCRIPTION:
Muscles to cause the weakened or paralyzed muscles to contract and produce a stepping motion of the legs. The FES stepping in this study will be done through a device called the RT600 FES Stepper (RT600).

ELIGIBILITY:
Inclusion Criteria:

* Male, Female, age 18-65, all ethnic groups
* Spinal Cord Injury, traumatic and non-traumatic
* C1-T12 neurological level
* ASIA class A-D
* Chronic injury > 6 months from the injury
* Visible motor response to FES stimulation (visible muscle contraction evoked with electrical stimulation)
* Subjects are medically stable, with no recent (1 month or less) inpatient admission for acute medical or surgical issues
* Subjects are able to comply with procedures and follow-up

Exclusion Criteria:

* Concurrent lower motor neuron disease such as peripheral neuropathy that would exclude lower extremity electrical excitability
* History of inability to tolerate electrical stimulation
* Cardiovascular disease as defined by previous myocardial infarction, unstable angina, requirement for anti platelet agents, congestive heart failure, or stroke NYHA Class III or IV, history of arrhythmia with hemodynamic instability
* Uncontrolled hypertension (resting systolic BP > 160mmHg or diastolic BP >100mmHg consistently)
* Presence of a pacemaker, an implanted defibrillator or certain other implanted electronic or metallic devices other than baclofen pumps
* Unstable long bone fractures of the lower extremities
* Presence of stage III or greater skin ulcerations that would preclude application of stimulating pads
* Malignancy
* History of epileptic seizures
* Women who are pregnant
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Fractures less than 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina L Sadowsky, MD, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FES Stepping
Started | 12
Completed | 10
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Groups:
- FES Stepping: FES Stepping, twice a week, for 8 weeks.
Arm/Group | FES Stepping
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor and Sensory Scores of the ASIA Impairment Scale (AIS)
Description: Change in motor, pin prick, and light touch score components of the ASIA Impairment scale (AIS) after 8 weeks of stepping FES in persons with spinal cord injury. The AIS evaluates motor and sensory function and comprises motor (min 0, max 100), pin prick (min 0, max 112), and light touch (min 0, max 112) scores. Higher scores represent better functional outcome.
  AIS Classificatrion:
  A = Complete: No motor or sensory function is preserved in the sacral segments S4-S5.
  B = Incomplete: Sensory but not motor function is preserved below the neurological level and includes the sacral segments S4-S5.
  C = Incomplete: Motor function is preserved below the neurological level, and more than half of key muscles below the neurological level have a muscle grade less than 3.
  D = Incomplete: Motor function is preserved below the neurological level, and at least half of key muscles below the neurological level have a muscle grade of 3 or more.
  E = Normal: motor and sensory function are normal.
Time Frame: Baseline, 8 weeks
Measure: Mean (Full Range); unit: scores on AIS Scale
Arm/Group | FES Stepping
Number analyzed (Participants) | 10
scores on AIS Scale
  Upper Extremity Motor Score | 1.0 [0 to 5]
  Lower Extremity Motor Score | 2.7 [-1.0 to 7]
  Light Touch | 2.4 [-2.0 to 9]
  Pin prick | -1.2 [-16.0 to 11.0]

2. Secondary Outcome: Change in Heart Rate
Description: Change in heart rate following 8 weeks of FES. Change in heart rate from baseline was computed from week 8 parameters.
Time Frame: Baseline, 8 weeks
Measure: Mean (Full Range); unit: beats per minute
Arm/Group | FES Stepping
Number analyzed (Participants) | 10
beats per minute | -3.3 [-18 to 6]

3. Secondary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure following 8 weeks. Change in systolic blood pressure from baseline was computed from week 8 parameters.
Time Frame: Baseline, 8 weeks
Measure: Mean (Full Range); unit: mmHg
Arm/Group | FES Stepping
Number analyzed (Participants) | 10
mmHg | 1.1 [-24 to 23]

4. Secondary Outcome: Change in Diastolic Plood Pressure
Description: Change in distolic blood pressure following 8 weeks. Change in diastolic blood pressure from baseline was computed from week 8 parameters.
Time Frame: Baseline, 8 weeks
Measure: Mean (Full Range); unit: mmHg
Arm/Group | FES Stepping
Number analyzed (Participants) | 10
mmHg | 1.8 [-14 to 22]

5. Secondary Outcome: Change in Rate of Perceived Exertion
Description: Change in rate of perceived exertion (RPE) following 8 weeks of FES. Change in rate of perceived exertion (RPE) from baseline was computed from week 8 parameters.
  The RPE scale is a 15 point scale ranging from 6 to 20 points. Higher scores indicate greater exertion.
Time Frame: Baseline, 8 weeks
Measure: Mean (Full Range); unit: scores on RPE scale
Arm/Group | FES Stepping
Number analyzed (Participants) | 10
scores on RPE scale | -0.64 [-3.0 to 1.0]

6. Secondary Outcome: Change in Vital Capacity
Description: Change in vital capacity following 8 weeks of FES. Change in vital capacity from baseline was computed from week 8 parameters.
Time Frame: Baseline, 8 weeks
Measure: Mean (Full Range); unit: litres
Arm/Group | FES Stepping
Number analyzed (Participants) | 10
litres | -0.29 [-0.97 to 0.56]

7. Secondary Outcome: Change in Peak Cough Flow
Description: Change in cough flow following 8 weeks of FES. Change in peak cough flow from baseline was computed from week 8 parameters.
Time Frame: Baseline, 8 weeks
Measure: Mean (Full Range); unit: liters/minute
Arm/Group | FES Stepping
Number analyzed (Participants) | 10
liters/minute | -6 [-110 to 100]

ADVERSE EVENTS:
Arm/Group | FES Stepping
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FES Stepping (N=12)
Ankle Swelling (X-ray negative for bone fracture or dislocation) (Musculoskeletal and connective tissue disorders) | 2 (2) — Reported swelling and bruise on medial aspect of ankle X-ray negative for bone fracture, dislocation Resume FES stepping by taking precautions by giving ankles more support: ace bandage wrapping; wear ankle supportive running shoes (high tops)
Lightheadedness (Cardiac disorders) | 3 (3) — FES was stopped. participant rested, and symptoms resolved. Did not affect continued participation in study
Increased tone in lower extremity (Musculoskeletal and connective tissue disorders) | 3 (3) — Increased tone did not interfere with FES stepping

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes